CLINICAL TRIAL: NCT05115422
Title: Feasibility and Acceptability of a Virtual 'Coping With Brain Fog' Intervention for Adolescents and Young Adults With Cancer
Brief Title: Feasibility and Acceptability of a Virtual 'Coping With Brain Fog' Intervention for Young Adults With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Collaborators: CancerCare Manitoba (Other)
Responsible Party: Principal Investigator, Sapna Oberoi, Pediatric Hematologist Oncologist, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AYABF2021P
Record Dates: First submitted 2021-10-16; First posted 2021-11-10 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Cancer; Cognitive Dysfunction; Cognitive Impairment; Adolescents; Young Adults
Keywords: Brain fog; Psychological Distress; Anxiety; Depression; Fatigue
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction; Mental Fatigue; Anxiety Disorders; Depression; Fatigue | interventions — Coping Skills

STUDY DESIGN:
Intervention Model Description: Pilot study of the virtual 'Coping with Brain Fog' intervention for AYAs with cancer living in Manitoba.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Coping with Brain Fog" intervention (Experimental)
  Interventions: Behavioral: 'Coping with Brain Fog' program

INTERVENTIONS:
Behavioral: 'Coping with Brain Fog' program — The proposed intervention is an 8-week 'Coping with Brain Fog' program for cancer survivors, adapted for AYAs with cancer, with one 90-minute group session per week. The intended group size for the program is 8-12 participants. The program was developed to be delivered in person, however for the purposes of this study it will be conducted in a virtual setting. The overall goals of the program are to educate participants about cancer-related brain fog and enhance their cognitive function and wellbeing. To accomplish this, the program is segmented into three main components: memory skills, task management, and psychological wellbeing. For each component, participants are systematically introduced to evidence-based strategies to cumulatively build a repertoire of cognitive tools designed to reduce the impact of cancer-related brain fog. The program uses a manual and participant materials that are copyrighted by Maximum Capacity Inc.

SUMMARY:
Cancer-related cognitive problems, also known as "brain fog", have a significant impact on patients with cancer and cancer survivors. Previous studies indicate that cancer and cancer treatments can negatively affect memory, attention and thinking abilities. Adolescents and young adults (AYAs) are individuals with a cancer diagnosis, who are currently between 18 to 40 years old. These individuals are especially vulnerable to brain fog symptoms due to the effect these symptoms have on their education, employment, health behaviors, mental health, and social relationships. There is a clear need for programming directed at brain fog symptoms among AYAs with cancer diagnoses. The 'Coping with Brain Fog' program, developed by Maximum Capacity Inc., is an eight-week group program that has been designed to educate patients about their brain fog symptoms and develop strategies to manage these symptoms. In this study the investigators will aim to determine the feasibility of adapting the 'Coping with Brain Fog' program to the virtual setting for AYAs with cancer during the COVID-19 pandemic. The investigators will also aim to explore the efficacy of the program on cognitive functioning and symptoms of anxiety, depression and fatigue. This study is an important step towards finding ways to treat brain fog symptoms in cancer patients, and could help guide future studies and programs.

DETAILED DESCRIPTION:
Background: Cancer-related cognitive deficits, also known as "brain fog", are a well-established morbidity among patients with cancer and cancer survivors. Associations between cancer or cancer treatment with difficulties in short-term and working memory, attention, processing speed, verbal fluency, and executive function have been previously described. Adolescents and young adults (AYA) are individuals who have had a cancer diagnosis and are currently between 18 to 40 years of age. Mitigating cognitive symptoms in the AYA population is especially important, as these cognitive symptoms affect education and employment, health behaviors, mental health, and social relationships. Further, as more AYAs with cancer survive their cancer and live into adulthood, improving their quality of life is even more vital. There is a clear need for programming directed at brain fog symptoms among AYAs with a cancer diagnosis.

Objective: The primary objective of this study is to determine the feasibility and acceptability/satisfaction of a virtual 'Coping with Brain Fog' intervention to AYAs with cancer during the COVID-19 pandemic. Secondary objectives of the study are to determine the preliminary effect of the intervention on the cognitive functioning and symptoms of distress (anxiety/depression/fatigue) of AYAs with cancer.

Methods: This prospective pilot study will involve an 8-week virtual "Coping with Brain Fog" program, with one 90-minutes session per week. The 'Coping with Brain Fog' program, developed by Maximum Capacity Inc., has been designed as an in-person group program to educate participants about brain fog and help them enhance their cognition and overall wellbeing. Sessions are designed to enhance memory, task management, and psychological wellbeing skills. Sessions will be delivered over Zoom in a group setting by a Master's-prepared registered social worker and AYA psychosocial oncology clinician at CancerCare Manitoba. Individuals who are between the ages of 18-40 and are (a) diagnosed with any type or stage of cancer, (b) seeking intervention for self-reported symptoms of brain fog (such as poor memory, mental slowness, or task insufficiency), and (c) currently living in Manitoba, Northwestern Ontario or Nunavut, will be eligible for this study. Before starting the intervention, the study participants will be sent a survey link to collect background patient information and measure self-reported cognitive function and symptoms of distress. The participants will also complete a post-intervention questionnaire to measure self-reported cognitive function, symptoms of distress, and satisfaction within one week of completing the intervention and at 6-8 weeks after the intervention. Semi-structured exit phone interviews will be conducted with the participants within two weeks of completing the intervention to collect their narrative feedback and experiences with the intervention.

Significance: This pilot project will help determine the feasibility and acceptability/satisfaction of a virtual 'Coping with Brain Fog' program and measure its preliminary effects on cognitive function and symptoms of distress among AYAs with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Diagnosed with any type or stage of cancer
* Seeking intervention for self-reported symptoms of brain fog (such as poor memory, mental slowness, or task insufficiency)
* Must be currently living in Manitoba, Nunavut or Northwest Ontario
* Must be able to attend eight virtual sessions of the 'Coping with Brain Fog' intervention
* Must have reliable access to the internet and the audio-visual platform Zoom
* Should also be able to read, speak and write English (as the sessions will be conducted in English)

Exclusion Criteria:

* Age younger than 18 or older than 40 years at the time of enrollment
* Must not have a previously diagnosed severe intellectual disability (self-reported by the participants)
* Should not be receiving any new interventions to enhance their cognitive function during the period of this study
* Must attend the first two sessions and should not miss two consecutive sessions (if a participant misses two consecutive sessions due to extenuating circumstances, they will be encouraged to withdraw from the group and be prioritized on the wait-list for the next brain fog group)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | Adherence will be assessed at the end of the 8-week intervention.
  The investigators will measure the adherence to the intervention by measuring attendance at the weekly sessions. The intervention will be considered feasible if 60% of participants do not miss the first two sessions and any two consecutive sessions.
Participant Satisfaction - Client Satisfaction Questionnaire | Participant Satisfaction will be measured at the end of the 8-week intervention.
  The participants' satisfaction with the program will be measured using The Client Satisfaction Questionnaire (CSQ), an 8-item self-report scale which will be administered at the end of the intervention to assess the participant satisfaction. Each item on this scale is scored from 1 to 4, generating a total score ranging from 8 to 32. A total score of 8-20 indicates low satisfaction, whereas total scores of 21-26 and 27-32 indicate medium and higher satisfaction, respectively.

SECONDARY OUTCOMES:
Perceived Cognitive Functioning - Functional Assessment of Cancer Therapy-Cognitive Function Scale | The investigators will measure perceived cognitive functioning before, one week after, and 6-8 weeks after the intervention.
  The investigators will measure perceived cognitive functioning before and after the intervention using the Functional Assessment of Cancer Therapy (FACT)-Cognitive Function Scale, a 37-item self-report scale, which will be administered to measure subscales of perceived cognitive impairments, impact of perceived cognitive impairments on quality of life, comments from others, and perceived cognitive abilities. Each item on the subscales is scored from 0 to 4, to generate a total score for each subsection. These subscale scores will be aggregated to give a final score between 0-20, with a higher score being associated with better quality of life.
Perceived Cognitive Functioning - Cancer Distress Scales for Adolescents and Young Adults | The investigators will measure perceived cognitive functioning before, one week after, and 6-8 weeks after the intervention.
  The investigators will measure perceived cognitive functioning before and after the intervention using the Cognitive component of the Cancer Distress Scales for Adolescents and Young Adults (CDS-AYA), an 8-item self-report scale, which will be administered before and at the end of the intervention to measure distress related to cognitive problems. Each item on this scale is scored from 0 to 3 to generate a total score between 0-24. Raw sum scores are transformed to a score from 0 (best) to 100 (worst), with a higher score reflecting more distress.
Symptoms of Distress and Fatigue - Anxiety | The investigators will measure symptoms of distress before, one week after, and 6-8 weeks after the intervention.
  The investigators will evaluate anxiety using the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Anxiety 8a, an 8-item self-report scale. Each item on the form is scored from 0 (never) to 5 (always). Scores on each item are summed to determine a raw score, which is converted to a standardized T-score with a mean of 50 and a standard deviation (SD) of 10, with a higher score reflecting greater anxiety.
Symptoms of Distress and Fatigue - Depression | The investigators will measure symptoms of distress before, one week after, and 6-8 weeks after the intervention.
  The investigators will evaluate depression using the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Depression 8b, an 8-item self-report scale. Each item on the form is scored from 0 (never) to 5 (always). Scores on each item are summed to determine a raw score, which is converted to a standardized T-score with a mean of 50 and a standard deviation (SD) of 10, with a higher score reflecting greater depression.
Symptoms of Distress and Fatigue - Fatigue | The investigators will measure symptoms of distress before, one week after, and 6-8 weeks after the intervention.
  The investigators will evaluate fatigue using the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Fatigue 8a, an 8-item self-report scale. Each item on the form is scored from 0 (not at all/never) to 5 (very much/always). Scores on each item are summed to determine a raw score, which is converted to a standardized T-score with a mean of 50 and a standard deviation (SD) of 10, with a higher score reflecting greater fatigue.
Participant experience with the program using semi-structured exit interview | Exit interviews will occur at the end of the 8-week intervention.
  The semi-structured interview conducted at the end of the intervention will explore participants' experience with the program and satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- CancerCare Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardy SJ, Krull KR, Wefel JS, Janelsins M. Cognitive Changes in Cancer Survivors. Am Soc Clin Oncol Educ Book. 2018 May 23;38:795-806. doi: 10.1200/EDBK_201179. PMID 30231372
- [Background] Jean-Pierre P, Winters PC, Ahles TA, Antoni M, Armstrong FD, Penedo F, Lipshultz SE, Miller TL, Fiscella K. Prevalence of self-reported memory problems in adult cancer survivors: a national cross-sectional study. J Oncol Pract. 2012 Jan;8(1):30-4. doi: 10.1200/JOP.2011.000231. Epub 2011 Nov 22. PMID 22548008
- [Background] Prasad PK, Hardy KK, Zhang N, Edelstein K, Srivastava D, Zeltzer L, Stovall M, Seibel NL, Leisenring W, Armstrong GT, Robison LL, Krull K. Psychosocial and Neurocognitive Outcomes in Adult Survivors of Adolescent and Early Young Adult Cancer: A Report From the Childhood Cancer Survivor Study. J Clin Oncol. 2015 Aug 10;33(23):2545-52. doi: 10.1200/JCO.2014.57.7528. Epub 2015 Jul 6. PMID 26150441
- [Background] McDougall GJ Jr, Oliver JS, Scogin F. Memory and cancer: a review of the literature. Arch Psychiatr Nurs. 2014 Jun;28(3):180-6. doi: 10.1016/j.apnu.2013.12.005. Epub 2014 Mar 22. PMID 24856270
- [Background] Ahles TA, Root JC, Ryan EL. Cancer- and cancer treatment-associated cognitive change: an update on the state of the science. J Clin Oncol. 2012 Oct 20;30(30):3675-86. doi: 10.1200/JCO.2012.43.0116. Epub 2012 Sep 24. PMID 23008308
- [Background] Barnett M, McDonnell G, DeRosa A, Schuler T, Philip E, Peterson L, Touza K, Jhanwar S, Atkinson TM, Ford JS. Psychosocial outcomes and interventions among cancer survivors diagnosed during adolescence and young adulthood (AYA): a systematic review. J Cancer Surviv. 2016 Oct;10(5):814-31. doi: 10.1007/s11764-016-0527-6. Epub 2016 Feb 26. PMID 26920873
- [Background] Perales MA, Drake EK, Pemmaraju N, Wood WA. Social Media and the Adolescent and Young Adult (AYA) Patient with Cancer. Curr Hematol Malig Rep. 2016 Dec;11(6):449-455. doi: 10.1007/s11899-016-0313-6. PMID 26893061
- [Background] Anderson C, Nichols HB. Trends in Late Mortality Among Adolescent and Young Adult Cancer Survivors. J Natl Cancer Inst. 2020 Oct 1;112(10):994-1002. doi: 10.1093/jnci/djaa014. PMID 32123906
- [Background] Miller KD, Fidler-Benaoudia M, Keegan TH, Hipp HS, Jemal A, Siegel RL. Cancer statistics for adolescents and young adults, 2020. CA Cancer J Clin. 2020 Nov;70(6):443-459. doi: 10.3322/caac.21637. Epub 2020 Sep 17. PMID 32940362
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Tsangaris E, D'Agostino N, Rae C, Breakey V, Klassen AF. Development and Psychometric Evaluation of the Cancer Distress Scales for Adolescent and Young Adults. J Adolesc Young Adult Oncol. 2019 Oct;8(5):566-580. doi: 10.1089/jayao.2019.0005. Epub 2019 Jul 8. PMID 31274372
- [Derived] Muthumuni D, Scott I, Chochinov HM, Mahar AL, Garland SN, Schulte F, Lambert P, Lix L, Garland A, Oberoi S. Feasibility and Acceptability of a Virtual "Coping with Brain Fog" Intervention for Improving Cognitive Functioning in Young Adults with Cancer. J Adolesc Young Adult Oncol. 2023 Oct;12(5):662-673. doi: 10.1089/jayao.2023.0022. Epub 2023 May 8. PMID 37158780
- See also: Related Info — http://www.maximumcapacity.org/
- See also: PROMIS Short Form v1.0 - Anxiety 8a — https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=147&Itemid=992
- See also: PROMIS Short Form v1.0 - Depression 8b — https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=157&Itemid=992
- See also: PROMIS Short Form v1.0 - Fatigue 8a — https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=161&Itemid=992